CLINICAL TRIAL: NCT07149090
Title: A Clinical Trial Evaluating the Efficacy and Safety of Lenvatinib, Nivolumab, and Chemotherapy in Metastatic Gastric Cancer With Malignant Ascites.
Brief Title: Lenvatinib in Combination With Nivolumab Plus Chemotherapy in Metastatic Gastric Cancer Patients With Malignant Ascites
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hyung-Don Kim, Assistant Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC2501
Record Dates: First submitted 2025-08-19; First posted 2025-08-29 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-08

CONDITIONS: STOMACH NEOPLASM; Gastric Cancer; Gastric Cancer Adenocarcinoma Metastatic
Keywords: Stomach Neoplasms; Gastric cancer; Lenvatinib; Advanced Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenvatinib+Nivolumab+Chemotherapy(Capecitabine+Oxaliplatin) (Experimental)
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Description: Lenvatinib: 12 mg (for body weight ≥ 60 kg) or 8 mg (for body weight < 60 kg) per oral once daily
  * Dose level 1: 8mg per oral once daily (for <60kg) 12mg per oral once daily (for ≥ 60kg)
  * Dose level 2: 4mg per oral once daily (for <60kg) 8mg per oral once daily (for ≥ 60kg) Nivolumab: 360 mg administered intravenously every 3 weeks Chemotherapy(Oxaliplatin+Capecitabine) every 3 weeks
  * Capecitabine 1000 mg/m² per oral twice daily on Days 1-14
  * Oxaliplatin 130 mg/m² administered intravenously on Day 1
  Other Names: Nivolumab+Chemotherapy(Capecitabine+Oxaliplatin)

SUMMARY:
To investigate efficacy and safety of lenvatinib in combination with nivolumab plus chemotherapy in gastric cancer patients with peritoneal metastasis and grade ≥ 2 ascites.

DETAILED DESCRIPTION:
Gastric cancer is the 4th leading cause of cancer-related mortality and the 5th most common malignancy worldwide. The past decade has seen significant progress in first-line systemic chemotherapy for patients with advanced gastric cancer. Immune checkpoint inhibitor (ICI)-based chemotherapy has become the standard first-line treatment since the demonstration of improved overall survival (OS) due to nivolumab plus chemotherapy in the Checkmate-649 study. Subsequent phase 3 trials have also demonstrated the positive impact of adding ICI to chemotherapy on survival. However, a proportion of patients still show poor survival outcomes with first-line ICI plus chemotherapy, highlighting an unmet need to improve treatment outcomes in such patients.

While patients with microsatellite instability (MSI)-high gastrointestinal cancers exhibit favorable outcomes with ICIs, MSI-high gastrointestinal cancers with peritoneal metastases and ascites exhibited highly unfavorable outcomes to ICI-based therapies. To this end, a research team analyzed the survival outcomes of gastric cancer patients treated with first-line nivolumab plus chemotherapy, finding that patients with peritoneal metastasis and grade ≥ 2 ascites had detrimental survival outcomes despite a high PD-L1 CPS (≥5). Ascites VEGF level was reportedly high in patients with a large amount of malignant ascites, supporting the concept that anti-VEGF therapies are promising for treating gastric cancer patients with peritoneal metastasis.

Lenvatinib is a potent multiple RTKi that selectively inhibits VEGF receptors, VEGFR1 (FLT1), VEGFR2 (KDR), VEGFR3 (FLT4), FGFR1-4, PDGFRα, c-KIT, and RET, which is approved for use in various cancer types, including hepatocellular carcinoma. Among known kinase inhibitors in clinical use, lenvatinib is one of the only inhibitors currently labeled with a mechanism of action as an inhibitor of not only VEGFRs but also FGFRs, both of which are currently believed to be very important for tumor angiogenesis.

It is hypothesized that the addition of lenvatinib to nivolumab plus chemotherapy in gastric cancer patients with peritoneal metastasis and grade ≥ 2 ascites could improve survival outcomes for these patients. A prospective phase Ib/II trial has been designed to investigate the efficacy and safety of lenvatinib in combination with nivolumab plus chemotherapy in gastric cancer patients with peritoneal metastasis and grade ≥ 2 ascites.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed pathologically proven metastatic, unresectable or recurrent gastric or gastroesophageal junction (GEJ) adenocarcinoma
2. Positive for peritoneal metastasis and grade ≥ 2 malignant ascites as confirmed by computed tomography (CT)
3. PD-L1 combined positive score of ≥5 based on the 28-8 assay
4. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations
5. Age > 19 years at time of study entry
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Life expectancy of > 4 months
8. Body weight > 30kg
9. No existing neuropathy
10. Adequate normal organ and marrow function as defined below:

    * Hemoglobin ≥9.0 g/dL
    * Absolute neutrophil count (ANC) 1.5 x (> 1500 per mm3)
    * Platelet count ≥100 (or 75) x 109/L (>75,000 per mm3)
    * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN)
    * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional ULN
    * Measured creatinine clearance (CL) > 40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance:
11. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre- menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.
12. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

1. Disease progression within 6 months after completion of adjuvant chemotherapy.
2. Participation in another clinical study with an investigational product during the last 2 weeks
3. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
4. Any concurrent chemotherapy, immunotherapy, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable
5. Major surgical procedure within 28 days prior to the first dose
6. Unable to take medication orally
7. Gastrointestinal bleeding
8. Impaired bowel absorption
9. History of allogenic organ transplantation
10. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events (AEs) or compromise the ability of the patient to give written informed consent
11. History of another primary malignancy except for

    * Malignancy treated with curative intent and with no known active disease ≥ 5 years before the first dose and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease
12. History of active primary immunodeficiency
13. Active infectious disease
14. Tuberculosis (based on clinical history, physical examination, radiographic findings, and TB testing in line with local practice)
15. Hepatitis B (known positive HBV surface antigen (HBsAg) result)
16. Hepatitis C (patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA)
17. Human immunodeficiency virus (positive HIV 1/2 antibodies)
18. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible.
19. Female patients who are pregnant or breastfeeding, as well as male or female patients of reproductive potential who are not willing to use effective contraception from the time of screening until 5 months following the final dose of lenvatinib.
20. Known allergy or hypersensitivity to the investigational drug or any of its components.
21. Patients with known deficiency of dihydropyrimidine dehydrogenase (DPD).
22. Patients with known hereditary problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1b part: Recommend phase 2 dose(RP2D) | At the end of Cycle 1 (each cycle is 21 days)
  Phase 1b part: will follow a traditional 3+3 dose-escalation design. Dose-limiting toxicities (DLTs) will be assessed after the first 3 subjects are enrolled. If no DLTs are observed among the initial 3 subjects, the dose level will be considered the recommended phase 2 dose (RP2D). If 1 of the initial 3 subjects experiences a DLT, 3 additional subjects will be enrolled at the same dose level (for a total of 6 subjects). If ≤1 of 6 subjects experience a DLT, the dose level will be defined as the RP2D. Up to 12 subjects may be enrolled in the Phase 1b part.
Phase II part: 6 month progression-free survival (PFS) rate | At 6 months
  6 month progression-free survival (PFS) rate

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No